CLINICAL TRIAL: NCT04604028
Title: A Phase II Trial of Combination of Oral Lenalidomide and Low-dose Cyclophosphamide for Patients With Antibiotics-unresponsive Extranodal Marginal Zone B-cell Lymphoma
Brief Title: Lenalidomide and Low-dose Cyclophosphamide for MALT Lymphoma
Acronym: LCMALT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202003096MIPC
Record Dates: First submitted 2020-09-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-09

CONDITIONS: Antibiotics-unresponsive MALT Lymphoma; Relapsed MALT Type Extranodal Marginal Zone B-Cell Lymphoma; Refractory Extranodal Marginal Zone B-Cell Lymphoma (MALT)
Keywords: Marginal zone B-cell lymphoma; Low-dose Cyclophosphamide; Lenalidomide
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide and low-dose cyclophosphamide (Experimental): Oral lenalidomide and low-dose cyclophosphamide (LC: lenalidomide [Leavdo®] 15 mg daily, day 1 to day 21; cyclophosphamide [Endoxan] 50 mg daily, day 1 to day 21; courses will be repeated every 28 days
  Interventions: Drug: Lenalidomide [Leavdo®]

INTERVENTIONS:
Drug: Lenalidomide [Leavdo®] — Complete remission and partial remission rate
  Other Names: Low-dose cyclophosphamide

SUMMARY:
Considering that lenalidomide and cyclophosphamide are found to have anti-tumor effects in MALT lymphoma, the investigators speculated that combined lenalidomide and low-dose cyclophosphamide can increase the overall response rate as well as dural time of tumor remission, and avoid alternative treatments, including radiotherapy or chemotherapy-related adverse effects in antibiotics-unresponsive, relapsed or refractory extranodal MALT lymphoma. Therefore, in this proposal, the investigators will design a prospective phase II study to evaluate the treatment efficacies of combination of oral lenalidomide and low-dose cyclophosphamide (LC: lenalidomide [Leavdo®] 15 mg daily, day 1 to day 21; cyclophosphamide [Endoxan] 50 mg daily, day 1 to day 21; courses will be repeated every 28 days) in patients with antibiotics-unresponsive, relapsed or refractory extranodal MALT lymphoma.

DETAILED DESCRIPTION:
[Background]: In addition to Helicobacter pylori-negative gastric marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (named as MALT lymphoma) (Sci Rep. 2017;7(1):14333), the investigators recently demonstrated that first-line antibiotics treatments can cure around 50% patients with stage IE/IIE1 extragastric MALT lymphoma (2018 ESMO poster discussion). However, the optimal management for antibiotics-unresponsive MALT lymphomas is not clearly defined.

[Rationale]: The investigators previously reported that thalidomide resulted in an overall response rate (ORR, including complete remission [CR] and partial remission [PR]) of 50% in 10 patients with antibiotics-unresponsive or chemotherapy-resistant MALT lymphoma. Lenalidomide (an immunomodulatory derivatives [IMiDs] of thalidomide) exhibits anti-angiogenic and immunomodulatory effects and has been proved efficacies in the treatment of multiple myeloma (MM). In the previous phase II study, single agent of lenalidomide resulted in ORR of 61.1% in 18 patients with MALT lymphoma. In addition to kill lymphoma cells, single low-dose cyclophosphamide, is an option for restoring immune response in patients with advanced cancer. The investigators also showed that low-dose cyclophosphamide (50 mg daily for 21 days, every 28 days) alone resulted in the ORR of 44.4 % in 9 patients with antibiotics-unresponsive MALT lymphoma. Previous studies also demonstrated that the addition of low-dose cyclophosphamide can overcome lenalidomide resistance in patients with MM.

[Hypotheses]: Considering that lenalidomide and cyclophosphamide are found to have anti-tumor effects in MALT lymphoma, the investigators speculated that combined lenalidomide and low-dose cyclophosphamide can increase the ORR rate as well as dural time of tumor remission, and avoid alternative treatments, including radiotherapy or chemotherapy-related adverse effects in antibiotics-unresponsive, relapsed or refractory extranodal MALT lymphoma.

[Methods]: Therefore, in this proposal, the investigators will design a prospective phase II study to evaluate the treatment efficacies of combination of oral lenalidomide and low-dose cyclophosphamide (LC: lenalidomide [Leavdo®] 15 mg daily, day 1 to day 21; cyclophosphamide [Endoxan] 50 mg daily, day 1 to day 21; courses will be repeated every 28 days) in patients with antibiotics-unresponsive, relapsed or refractory extranodal MALT lymphoma. The primary endpoint of this current study is ORR, and the second endpoint is adverse effect. The investigators will enroll 21 patients with antibiotics-unresponsive, relapsed or refractory MALT lymphoma based on the Simon minimax two-stage design.

The translational studies, including predictive markers and immunological profiles (BAFF-related canonical and non-canonical NF-κB signaling molecules, and immune-related molecules markers) will be included in the second points. The investigators will further assess immune-related molecules of nucleated cells of whole blood using flow cytometry, and analyze serum BAFF and cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified diagnosis of MALT lymphoma arising at any extranodal site
2. Diseases of extranodal MALT lymphoma 2.1 It does not initially respond to antibiotics or 2.2 It is refractory to or in first or greater relapse after prior radiotherapy and/ or chemotherapy and/or immunotherapy
3. Measurable or non-measurable lesions where the response is nevertheless evaluable by non-imaging means (e.g., gastric or bone marrow infiltrations)
4. Ann Arbor Stage I-IV
5. ECOG performance status of 0, 1 or 2
6. Age ≥ 18 years
7. Life expectancy of at least 3 months
8. Adequate haematological status: ANC (absolute neutrophil count [segmented + bands]) ≥1.0 x 109/L, platelet count ≥ 75 x 109/L , haemoglobin ≥8 g/dL.
9. Adequate cardiac, renal and liver function tests (serum creatinine < 2.0 mg/dl, ALT or AST < 2.5 x upper limit of normal range, alkaline phosphatase < 2.5 x upper limit of normal range, serum bilirubin < 2.0 mg/dl)
10. Patient must be willing and able to comply with the protocol for the entire study duration
11. Female patients of childbearing potential must agree to use, and be able to comply with, effective contraception and agree to have medically supervised pregnancy tests prior to starting the study treatment and during therapy
12. Male patients must agree to always use a condom during any sexual contact with females of reproductive potential and agree to not donate sperm while taking lenalidomide
13. Patient must agree to abstain from donating blood while taking study drug therapy
14. Patient must agree not to share study medication with another person and to return all unused study drug to the investigator

Exclusion Criteria:

1. Lymphoma histology other than MALT lymphoma or MALT lymphoma with a diffuse large cell lymphoma ("high grade lymphoma") component
2. Use of any investigational agent within 28 days prior to initiation of treatment
3. History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix or carcinoma in situ of the breast within the last 5 years unless in complete remission since at least 3 years
4. Dependency on red blood cell and/or platelet transfusions
5. Evidence of central nervous system involvement
6. A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
7. Severe peripheral polyneuropathy
8. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months and/or long QT-syndrome
9. HIV seropositivity
10. Presence of active opportunistic infections
11. Pregnancy or lactation
12. Uncontrolled diabetes mellitus
13. Pre-existing thromboembolic conditions at study entry
14. Known hypersensitivity to thalidomide or lenalidomide antibiotics
15. History of intolerance or hypersensitivity to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 1 year
  Included complete remission [CR] and partial remission [PR]

SECONDARY OUTCOMES:
Adverse Events assessments | 1 year
  Treatment-emergent adverse events (AEs) incidence, severity and relationship to study. treatment
Biomakers | 1 year
  Predict the response of combination of lenalidomide and cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hsin Kuo, M.D.,Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No